CLINICAL TRIAL: NCT05951114
Title: The Development of Post-operative Respiratory Muscle Dysfunction in Neurosurgical Patients
Brief Title: Post-neurosurgical Respiratory Muscle Dysfunction
Status: Recruiting | Type: Observational
Sponsor: Beijing Sanbo Brain Hospital (Other)
Responsible Party: Principal Investigator, Zhonghua Shi, MD, PhD, Deputy president of the department ICU, Beijing Sanbo Brain Hospital
Other Study IDs: HP2023-28-508001
Record Dates: First submitted 2023-06-08; First posted 2023-07-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-04

CONDITIONS: Diaphragm Issues; Neurosurgery; Pulmonary Complication
Keywords: Neurosurgery; Respiratory muscle dysfunction; Diaphragm; Expiratory muscle; Post operative pulmonary complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample will be collected based on clinical routine, and IL-6, IL-10, TNFα, NSE
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with diaphragm weakness: Diaphragm weakness will be defined as thickening fraction <=20 % at the time of extubation
  Interventions: Diagnostic Test: Maximum inspiratory/Expiratory manoeuvre for patients can follow the order
- Patients without diaphragm weakness: Diaphragm thickening fraction >20 % at the time of extubation
  Interventions: Diagnostic Test: Maximum inspiratory/Expiratory manoeuvre for patients can follow the order

INTERVENTIONS:
Diagnostic Test: Maximum inspiratory/Expiratory manoeuvre for patients can follow the order — Bedside ultrasound will be performed for each patient at the time before, after surgery, before and after extubation, and at the time of ICU discharge, under the end-expiratory occlusion, maximum inspiratory, and/or expiratory manoeuvre
  Other Names: End-expiratory occlusion in patients with endotracheal tube in situ

SUMMARY:
Respiratory muscle dysfunction may contribute to the development of postoperative pulmonary complications. However, it prevalence in patients receiving neurosurgery is largely unknown. Therefore, in present study, respiratory muscle function (measured by the ultrasound) and their correlation with the post-operative pulmonary complications will be analyzed.

DETAILED DESCRIPTION:
Postoperative pulmonary complications is common in patients receiving neurosurgery, and is associated with hospitalization cost and mortality. Respiratory muscle dysfunction is an important cause postoperative pulmonary complications, however, it's prevalence in patients receiving neurosurgery is unclear.

The diaphragm and abdominal expiratory muscles are the main inspiratory and expiratory driving muscles. Ultrasound can assess the function and morphology of these muscles invasively and in realtime. Studies has demonstrated their feasibility and repeatability in realtime monitoring of respiratory muscles.

In this study, our primary aim is to assess the respiratory muscle function after neurosurgery, and the correlation between diaphragm and expiratory muscle function. Our secondary aims including the correlation between the brain injury and the respiratory muscle function, and the impact of post-operative respiratory muscle dysfunction on the pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* First elective operation during hospitalization
* ASA<3

Exclusion Criteria:

* Brain stem and spinal spine lesions
* Preoperative chest imaging findings were abnormal
* Mechanical ventilation was required before surgery
* Clinical or radiological evidence of preoperative misaspiration
* History of neurosurgery in the last 6 months
* A history of neuromuscular disease
* BMI≥35kg/m2
* Pregnant women
* Skin lesions detected by ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving elective surgery
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of diaphragm dysfunction after neurosurgery | Within 24 hours after the completion of surgery
  The diaphragm dysfunction is defined as the thickening fraction < 20% under the maximum inspiration

SECONDARY OUTCOMES:
The correlation between the level of NSE and the diaphragm function | Within 24 hours after the completion of surgery
  The level of NSE is measured in the blood sample within 24 hours after surgery
The correlation between the level of inflammation maker ILs and the diaphragm function | Within 24 hours after the completion of surgery
  The level of ILs are measured in the blood sample within 24 hours after surgery
The correlation between the level of inflammation maker TNF-alpha and the diaphragm function | Within 24 hours after the completion of surgery
  The level of TNF-alpha is measured in the blood sample within 24 hours after surgery
The thickening fraction of expiratory muscles after surgery | Within 24 hours after the completion of surgery
  the thickening fraction of expiratory muscle is measured under the maximum expiration maneuver
The incidence of postoperative pulmonary complication | Through study completion, an average of 1 month
  The postoperative pulmonary complication is defined as when patient has developed one or more complications including pneumonia, atelectasis, pulmonary edema, pulmonary embolism, or respiratory failure
The length of hospital stay | Through study completion, an average of 1 month
  The length of hospital stay is counted by day
The length of ICU stay | Through study completion, an average of 1 month
  The length of ICU stay is counted by day
Duration of mechanical ventilation | Through study completion, an average of 1 month
  The duration of mechanical ventilation is counted by hours
Hospital mortality | Through study completion, an average of 1 month
  The hospital mortality is recorded at the time of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Zhonghua Shi, PhD, Principal Investigator — Capital Medical University
Locations (1):
- Beijing Sanbo Brain Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shi ZH, de Vries H, de Grooth HJ, Jonkman AH, Zhang Y, Haaksma M, van de Ven PM, de Man AAME, Girbes A, Tuinman PR, Zhou JX, Ottenheijm C, Heunks L. Changes in Respiratory Muscle Thickness during Mechanical Ventilation: Focus on Expiratory Muscles. Anesthesiology. 2021 May 1;134(5):748-759. doi: 10.1097/ALN.0000000000003736. PMID 33711154
- [Background] Shi ZH, Jonkman A, de Vries H, Jansen D, Ottenheijm C, Girbes A, Spoelstra-de Man A, Zhou JX, Brochard L, Heunks L. Expiratory muscle dysfunction in critically ill patients: towards improved understanding. Intensive Care Med. 2019 Aug;45(8):1061-1071. doi: 10.1007/s00134-019-05664-4. Epub 2019 Jun 24. PMID 31236639
- [Background] Tuinman PR, Jonkman AH, Dres M, Shi ZH, Goligher EC, Goffi A, de Korte C, Demoule A, Heunks L. Respiratory muscle ultrasonography: methodology, basic and advanced principles and clinical applications in ICU and ED patients-a narrative review. Intensive Care Med. 2020 Apr;46(4):594-605. doi: 10.1007/s00134-019-05892-8. Epub 2020 Jan 14. PMID 31938825